CLINICAL TRIAL: NCT05733962
Title: Multicentric Before/After Study to Assess the Efficacy and Safety of DBL-4pen Mobile Application on Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Evaluation of the Efficacy and Safety of DBL-4pen Mobile Application in Patients With Type 2 Diabetes
Acronym: SERENIT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diabeloop (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCB 2022-A00478-35
Record Dates: First submitted 2022-05-02; First posted 2023-02-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: regulation algorithm; Diabetes; Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: interventional single-arm open-label before/after multicentric national study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the device DBL-4pen (Experimental): After a 14-day baseline period during which the patient will use a Dexcom G6 Continuous Glucose Monitoring (CGM) and his current therapy (multiple daily injection), the patient will start a 42-day treatment period with the DBL-4pen system followed by an optional 42-day extension period.
  Interventions: Device: Use of the device DBL-4pen

INTERVENTIONS:
Device: Use of the device DBL-4pen — During the treatment period, the patient will use
  * the DBL-4pen device (consisting of a software hosting the Diabeloop algorithm installed on a smartphone)
  * the associated device #1: Dexcom G6, Continuous Glucose Monitoring (CGM)
  * the associated device #2: Two Mallya caps for their rapid- and long-acting insulin pens.
  The regulation algorithm hosted by DBL-4pen software recommends insulin doses to be administrated by the patient.

SUMMARY:
This study conducted in 40 adults living with type 2 diabetes is an interventional single-arm open-label before/after multicentric national study conducted as a clinical investigation according to the law EU 2017/745 art. 62.

After a 14-day baseline period during which the patient will use a Dexcom G6 Continuous Glucose Monitoring (CGM) and his current therapy (multiple daily injection), the patient will start a 42-day treatment period during which he will use the DBL-4pen application and two Mallya connected caps, in addition to the Dexcom G6 CGM. An optional 6-week extension period with treatment will be proposed to patients agreeing to pursue the use of DBL-4pen application.

The main objective is to evaluate the safety and efficacy of the DBL-4pen system for 6 weeks in patients with type 2 diabetes.

Data related to efficacy of DBL-4pen, global safety of DBL-4pen, compliance with recommended insulin injections, satisfaction with the system and quality of life will be collected.

The study is completed when all patients have their "end of study" file completed in the electronic Case Report Form (eCRF).

DETAILED DESCRIPTION:
This study conducted in 40 adults living with type 2 diabetes is an interventional single-arm open-label before/after multicentric national study conducted as a clinical investigation according to the law EU 2017/745 art. 62.

The study periods are as follows:

* 2 weeks of baseline period at home will be performed. During this baseline period, all patients will use their current therapy (MDI). In addition to their standard treatment, all patients will receive a Dexcom G6 and a smartphone. During this study period, the smartphone will be used to install the Dexcom G6 application in order to collect the glycemia data. The patients will make equivalent therapeutic decisions based on the values of the CGM used in the study (Dexcom G6) as if using their usual CGM.
* Followed by a 6-week treatment period: the patients will install the DBL-4pen application on the smartphone provided for the study with help of the research team and they will receive two Mallya caps for their insulin pens.
* Followed by an optional 6-week extension period with treatment for patients agreeing to pursue the use of the DBL-4pen system.

For each patient, a comparison will be made first between treatment and baseline periods and second between extension and baseline periods. In addition, a comparison of treatment vs extension periods will also be performed. Each patient will be his / her own control.

Visit 1: Inclusion and start of baseline phase for a duration of 2 weeks The investigator collects the dated and signed informed consent forms of patients who meet all inclusion and non-inclusion criteria.

Blood HbA1c test is performed in routine between one month before the V1 Visit and V1. If there is no routine HbA1c sampling during this period, the investigator will prescribe a study specific HbA1c blood test.

All patients are equipped with a Dexcom G6 CGM (instead of their usual CGM) and receive a smartphone on which they will install the Dexcom G6 application in order to collect interstitial glucose data. Patients will also be trained in the use of these devices by the medical team. Patients keep their current treatment (MDI) for the first phase of the study which will last two weeks. CGM parameters (such as alarms and alerts) will be matched with their usual treatment and patients will be asked to make equivalent therapeutic decisions based on the values of Dexcom G6 CGM as if using their usual CGM. In addition, for patients accustomed to using an interstitial glucose data visualization platform, the possibility of using Dexcom Clarity will be mentioned.

The site team will ensure and confirm the capacity of the patient to daily manage his Dexcom G6.

Visit 2 : V1 + 2 weeks (± 2 days) : End of baseline and start of the main treatment period The patient will install the investigational application DBL-4pen on the smartphone provided for the study and will be equipped with the Mallya caps and trained.

The site team will ensure and confirm the capacity of the patient to daily manage his DBL-4pen System and realize the device setting initialization.

The patient is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQs for satisfaction with his / her current treatment (see section 8.4 Secondary endpoints for more details on the questionnaires).

The qualified site staff reviews the patient's glucose control via Yourloops (a data visualization platform) and ensures the system is working as expected.

Visit 3 : V2 + 3 days (± 2 days): Phone call The qualified site staff review patient's glucose control via Yourloops at least twice a day during the first 3 days after the beginning of treatment.

Three days after installation of the DBL-4pen system, patients will be contacted by the qualified site staff to discuss its glycemic control and to adjust the system's parameters or patient's training if necessary. All related events are collected via eCRF.

Visit 4 : V2 + 3 weeks (± 2 days): Optional phone call After having reviewed the patient's glucose control via Yourloops, the medical staff will contact the patient after 3 weeks of using the DBL-4pen system if they consider that some adjustments are needed. More specifically, the medical staff will analyze the glycemic data with regard to the degree of use of the application by the patient and compliance with the recommendations. During this visit, adjustments in system settings or in its use by the patient (qualitatively and/or quantitatively) could be performed. If the medical staff finds that the glycemic control is stable, this visit will not take place.

Visit 5: V2 + 6 weeks (± 2 days) : End of the main treatment period - Start of extension (optional) The patient equipped with the DBL-4pen System can continue with the 6-week extension phase. During this visit, adjustments in system settings could be performed and recommendations, in particular on the use of the application by the patient, can be made.

The patient is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQs for satisfaction with DBL4-pen.

If they refuse to participate in the extension, the patients leave the study and the material is returned to the investigation site.

Visit 6: V5 + 6 weeks (± 2 days): End of study visit The patient is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQs for satisfaction with the system.

Blood HbA1c test is performed. The material is returned to the investigation site.

Contact by phone calls or additional visits are allowed during the study. They might be useful to discuss treatments, system parameters and adverse events. These additional visits can be initiated by the medical staff or by the patient. In addition, if the medical staff deems it necessary, the visits initially planned by telephone can be organized on site.

The main objective is to evaluate the safety and efficacy of the DBL-4pen system for 6 weeks in patients with type 2 diabetes. Analysis will be made between the 6-week treatment period versus the 2-week baseline period.

The secondary objectives of this study are to:

* assess the efficacy of DBL-4pen
* assess the global safety of DBL-4pen
* assess the compliance with recommended insulin injections
* assess the quality of life and satisfaction and adherence of subjects to the system

ELIGIBILITY:
Inclusion criteria:

Device-related inclusion criteria:

* Patients under basal-bolus scheme for type 2 diabetes
* Patients aged ≥ 18 years old
* Patients using rapid-acting analog and long-acting analog that are compatible with Mallya cap (Lispro, Detemir, Aspart, Glargine, Glulisine) with a stable insulin therapy regimen for at least the past 90 days (no modification of the number of injections and no more than 10% variation of the total daily dose)
* Patients using insulin with a concentration 100 U/mL

Study-specific inclusion criteria:

* No significant modification of diabetes treatment during the 3 months before inclusion (i.e., no introduction or removal of any pharmacological treatment, and no education training during this period), except for a possible modification for an equivalent insulin compatible with Mallya at least 15 days before inclusion
* Patients having an HbA1c ≤ 10%
* Patients who agree to use Dexcom G6 as CGM
* Patients living in an area covered by phone network
* Patients must be affiliated to any kind of social security
* Patients must be able to speak and be literate in French
* Non-isolated patients, not living alone, or having a "resource" person living nearby and having a telephone and the key of his home
* Having signed the free and informed consent form
* Subject equipped with a CGM for at least the past 90 days

Non-inclusion criteria

Device-related non-inclusion criteria

* Patients with Total Daily Dose (TDD) < 10 U
* Patients suffering from a serious illness or undergoing treatment that might significantly impair diabetes physiology, i.e. glucose-insulin interactions, that might interfere with the medical device (for example irregular treatment by steroids).
* Patients with severe uncorrected hearing impairment and/or severe uncorrected proble- ms of visual acuity.
* Patients unable to understand and perform instructions provided by Diabeloop SA.
* Patients who are unwilling or unable to maintain contact with the healthcare professional.
* Use of any insulin that is not 100U/mL rapid-acting insulin analog, 100U/mL long-acting insulin analog.

Study-specific non-inclusion criteria:

* Patients with type 1 diabetes
* Patients not feeling hypoglycemia (hypoglycemia unawareness)
* Patients who had an episode of severe hypoglycemia or a hypoglycemic coma in the past year while being equipped with any glucose sensor
* Patients not accepting to stay in France during the study
* Pregnant woman (verified by urine HCG pregnancy test for any woman wishing to participate in the protocol and of childbearing age < 60 year) or woman of childbearing potential in the absence of an effective method of contraception or if she does not agree to continue using contraception for the duration of the study
* Subjects under legal protection (guardianship, curatorship)
* Patients whose pancreas has been removed or is not functioning altogether
* Patients with islet/pancreas transplants.
* Patients with severely altered renal function (creatinine clearance <30 mL/min).
* Patients on dialysis
* Critically ill patients
* Any other physical or psychological disease, or medication likely to interfere with the conduct of the study and interpretation of the study results as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in 70 - 180 mg/dL glycemic range | 56 days
  Impact of the use of DBL-4pen on the time spent in the target 70-180 mg/dL during the main treatment period compared to baseline, in percentage.

SECONDARY OUTCOMES:
Percentage of time spent in specific glycemic ranges | 98 days
  Impact of the use of DBL-4pen on the time spent:
  * < 54 mg/dL
  * 54-69 mg/dL
  * < 70 mg/dL
  * 70-140 mg/dL
  * 70-180 mg/dL (for extension period)
  * > 180 mg/dL
  * 181-250 mg/dL
  * > 250 mg/dL
  during the main treatment period compared to baseline, and during the extension period compared to baseline, in percentage.
Mean CGM glycemia | 98 days
  Impact of the use of DBL-4pen on mean CGM records during the main treatment period compared to baseline, and during the extension period compared to baseline.
Variability of the glucose level | 98 days
  Impact of the use of DBL-4pen on the variability of the glucose level measured by the glycemic variation coefficient (CV) and Standard Deviation (SD) intra patient during the main treatment period compared to baseline, and during the extension period compared to baseline.
Glucose management indicator (GMI) | 98 days
  Impact of the use of DBL-4pen on the Glucose management indicator (GMI) during the main treatment period compared to baseline, and during the extension period compared to baseline. The formula used to calculate GMI is: GMI(%) = 3.31 + 0.02392 x [mean glucose in mg/dL].
Evolution of HbA1c for patients accepting the extension phase | 98 days
  Impact of the use of DBL-4pen on the evolution of HbA1c measured at baseline and after the extension period.
Incidence of severe hypoglycemia | 98 days
  Severe hypoglycemia is defined as hypoglycemia requiring third-party intervention OR with loss of consciousness OR involving hospitalization.
  The number of patients with severe hypoglycemia (and percentage) and the number of hypoglycemia events per week will be described overall and per study period.
Incidence of severe hyperglycemia | 98 days
  Severe hyperglycemia is defined as hyperglycemia with occurrence of ketoacidosis above 3 mmol/L OR involving hospitalization. The number of events per week, the number of patients with at least one episode (and percentage) will be described per study period and overall.
Number of adverse events, adverse device effects, serious adverse events, serious adverse device effects, unanticipated serious adverse device effects | 98 days
  The number of events, number of patients with at least one event (and percentage) will be described for the following type of adverse events:
  * Adverse Events (AEs)
  * Serious Adverse Events (SAEs)
  * Adverse Device Effects (ADEs)
  * Serious adverse Device Effects (SADEs)
  * Unanticipated Serious adverse Device Effects (USADEs)
Difference between the number of boluses recommended by the application and the number of boluses administered by the patient | 98 days
  The number of boluses recommended, administered per patient and the difference will be described per day for treatment and extension period. A recommended bolus is defined as an alert corresponding to a bolus recommendation (correction bolus and meal bolus recommendations).
  The potential factors associated with the difference between the number of boluses recommended by the application and administered by the patient will be investigated.
Difference between recommended and administered insulin dose | 98 days
  The total insulin dose per day and per patient will be described as a continuous parameter for treatment and extension period for recommended insulin and administered insulin. The difference between recommended and administered insulin dose will be described as absolute value and as the percentage of the recommended dose.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire total score | 98 days
  The Hypoglycemia Fear Survey (HFS) II questionnaire consists of 33 items. The HFS II score has a minimum of 0 and a maximum of 132. The higher the score, the more the patient fears hypoglycemia. The total score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire - Behaviour scale | 98 days
  The 15 items in Hypoglycemia Fear Survey (HFS-B) Behavior scale measure behaviors aimed at avoiding hypoglycemia and its possible negative consequences. The HFS-B score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared. The score has a minimum of 0 and a maximum of 60. The higher the score, the more the patient fears hypoglycemia.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire - Worrieness scale | 98 days
  The 18 items in Hypoglycemia Fear Survey (HFS-W) Worriedness scale measure various aspects relating to hypoglycemic episodes that provoke anxiety. The HFS-W score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared.
  The score has a minimum of 0 and a maximum of 72. The higher the score, the more the patient fears hypoglycemia.
Scoring of Diabetes Distress Scale (DDS) | 98 days
  The 17 items of DDS will be described both as continuous and categorical variables at baseline, treatment and extension period. Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem". Average scores will be computed and described for the four critical dimensions of distress: emotional burden, regimen distress, interpersonal distress and physician distress. The minimum and maximum scores will be 1 and 6, respectively.
  The evolution in DDS average score will be compared.The change in DDS will be evaluated between treatment and baseline period and between extension and baseline period.
Diabetes Treatment Satisfaction (DTSQs) Questionnaire items | 98 days
  The 8 DTSQ questionnaire items will be described as qualitative and quantitative outcomes at baseline, treatment and extension period. The minimum and maximum scores per item are 0 and 6, respectively. The higher the score, the more satisfied the patient is with the treatment.
  The evolution in score will be compared.
Scoring of Diabetes Treatment Satisfaction (DTSQs) Questionnaire | 98 days
  The DTSQ score is the sum of the 8 questionnaire items. It has a minimum of zero and a maximum of 36. The higher the score, the more satisfied the patient is with the treatment.
  DTSQ score will be described as continuous parameters at baseline, treatment and extension period.
  The evolution in score will be compared. The evolution in score will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves BENHAMOU, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble, Grenoble
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU Toulouse - Hôpital de Rangueil, Toulouse